CLINICAL TRIAL: NCT03819374
Title: Improving HIV/Tuberculosis Outcomes in Irkutsk
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Scientific Center for Family Health and Human Reproduction Problems, Russia (Other Government)
Responsible Party: Principal Investigator, Scott Heysell, MD, Associate Professor of Medicine, University of Virginia
Other Study IDs: 20451; R01DA044137 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis; HIV Infections; Substance Use
MeSH Terms: conditions — Tuberculosis; HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to examine the prospective influence of substance use patterns on HIV/tuberculosis adherence, pharmacokinetics and disease progression while developing novel methods for early detection and correction of these mechanisms of treatment failure in Irkutsk. At the University of Virginia, the investigators have considerable research experience with vulnerable HIV populations and have adapted mobile phone methods for data collection of adherence, substance use, and study retention. The investigators have also begun development of colorimetric methods for pharmacokinetic monitoring that utilizes urine which may be suitable as a non-invasive sample for the unique environmental factors affecting HIV patients in Irkutsk, namely geographic remoteness and concurrent substance use

DETAILED DESCRIPTION:
Subjects will be recruited at the Irkutsk Clinical Tuberculosis Hospital by trained research staff. Potential subjects are frequently diagnosed with HIV during their presentation with tuberculosis (TB) and treatment for TB begins prior to initiation of antiretrovirals for HIV. Hospital clinicians will notify research staff of potential subjects that are HIV infected, being treated for TB, have a history of substance use, and awaiting antiretroviral initiation. Prior to consent, potential subjects will be asked if they are willing to use a mobile phone as part of a research study. All subjects are consented in a private examination room by research staff. All enrolled subjects at each of the study sites are assigned individual participant identification (ID) numbers that are used for all subsequent case report forms and database.

Baseline characteristics and routine hospital laboratory data will be collected by the research staff from structured interview and review of hospital chart including demographics (age, sex, country/region of origin), CD4+ cell count and HIV viral load on admission to hospital (routine flow cytometry and Roche Amplicor version 1.5 for HIV-1 RNA levels- lower limit of detection 50 copies/mL), medical comorbidities other than HIV (diabetes, chronic kidney disease, hepatitis C or other known liver disease), and prior TB history, and anatomic site of current TB disease. Researchers will also compile a detailed substance use history and complete the HIV related quality of life survey, the Functional Assessment HIV Infection, that has been validated in the Russian setting.

Over the first 7 days of enrollment during hospitalization, the subject will receive education on the functionality of the smart phone including a short proficiency test that must be passed in order to have the mHealth application downloaded on their smartphone. In the rare instance that a subject does not own a smartphone, the study will issue a smartphone to the subject along with the dataplan. During that education period, the subject and the trained researcher will set-up the coding schema for the messages the subjects will later be texted. A preset coding schema will be available or the subject can individualize their messages with the researcher. If necessary, the researcher will explain the details of the smartphone "ownership" and data plan during the study period, how the data plan will be reissued each month, and if necessary, how the phone will be requested to be given back to the study staff after 6 months. The researchers acknowledge that some phones will not be retrieved, particularly in those subjects that die or experience permanent treatment cessation. In the situation where a subject cannot be confirmed as having died but does not present for one of the follow-up specimen collection procedures, the mHealth application will continue to send messages for the 6 month period that could record ongoing medication adherence (or non-adherence) and substance use.

Following the procedures that occur within the first 7 days of enrollment, phlebotomy and urine collection for pharmacokinetic testing will be scheduled to be performed after the patient has initiated anti-TB and antiretroviral treatment (between 2 and 8 weeks after hospitalization). Subjects remain in the hospital during this period per current clinical protocol/ standards of care. On the day of phlebotomy and urine collection, all medication will be directly administered and observed by nursing staff in the fasting state. All medications are given as a morning dose, and then venous blood samples are collected at 1, 2, 6 and optionally at 8 hours after the observed dose. A maximum of 5 ml will be obtained at each draw as up to 4 different anti-TB drugs will be required to be assayed by conventional chromatography methods. Blood will be immediately centrifuged onsite at the hospital and serum stored in sealed screw-cap tubes at -80 degrees Centigrade with the subject's participant ID number, sample ID number and study visit/time of blood draw. Batched serum specimens will be tested at the Scientific Centre in Irkutsk by chromatography/mass spectrometry. The sampling intervals allow for accurate estimates of the peak drug concentration (Cmax) and the area under the concentration curve (AUC), the two most important pharmacokinetic determinants of efficacy for the medications sampled. Urine will be collected for 24 hours (and labeled/stored as above) on the same day starting as soon as possible after medication administration. Urine will also be tested at the Scientific Centre in batch using the colorimetric assays. The first full 24 hour of urine drug concentration testing compared to the serum studies will allow adequate comparison of urinary kinetics to estimate the Cmax values from the timing of follow-up samples collected at 2 and 6 months after enrollment.

Following discharge from the hospital, subjects will be monitored for adherence by the daily messaging of the mobile health (mHealth) application and by monthly via medication refill reports from the TB Control Program. Subjects will be asked to return for follow-up visits at 2 and 6 months after enrollment. The site of follow-up will be arranged to be the TB clinic closest to where the patient resides or the clinic of the patient's request. Using the mHealth application, subjects will be texted the date, time and location of their study follow-up and the request to confirm yes/no that they will attend. Subjects unable to follow-up will be offered another time and location for follow-up, and if unable to be reached by text, then contacted using the alternative phone number(s) provided at enrollment.

At the follow-up visits researchers will administer a short symptom screening/ examination, a structured interview on substance use and medication recall assessment, then observe the subject taking their medications. During the 3-6 hours after medication administration the subject will have urine collected twice. If the subject does not have medication on hand, then another opportunity for follow-up will be arranged including the possibility of sample collection at the subject's residence. These follow-up urine specimens will not be frequent enough to calculate a full AUC, but rather an estimate of the Cmax value which we hypothesize to be most affected by patterns of substance use (alcohol and heroin).

At the completion of study procedures, an optional focus group discussion will be conducted among 30 randomly selected and gender balanced subjects to assess the feasibility of using mHealth application beyond that as a research tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-64 years of age
* HIV infected (confirmed by medical chart review)
* Initiating TB treatment (with anti-TB medicine)
* Initiating HIV treatment (with antiretroviral medicine)
* History of any substance use (confirmed by medical chart review)
* Primary residence in Irkutsk City, Russian Federation

Exclusion Criteria:

* Unable or unwilling to operate a smartphone
* Pregnant at time of enrollment per lab results (urine or serum) from Medical Record
* Prisoners Cognitively unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected adults initiating anti-TB and antiretroviral therapy over the course of 1 year at Irkutsk Regional TB Hospital with a history of substance use will undergo prospective adherence and substance use data collection facilitated by a population-adapted smart phone application, to assess the impact of this technology on medication adherence.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Nonadherence as measured by clinic attendance, pharmacy refill and daily adherence response to the mHealth app will be more frequent in participants with ongoing substance use. | At 12 months from enrollment nonadherence will be compared among those with a without ongoing substance use
  Participants will be assessed for measurements of adherence by clinic attendance, pharmacy refill at each study visit. Antiretroviral and anti-tuberculosis medication adherence is also questioned daily through the mHealth application. Additionally, a trans-renal DNA assay be measured at baseline and subsequent study visits to detect the presence of M. tuberculosis fragments in the urine.

SECONDARY OUTCOMES:
Correlation of serum mass spectrometry to urine colorimetry for AUC of anti-tuberculosis drugs | 6 months after enrollment completed
  Urine colorimetry will be compared to conventional serum mass spectrometry for kinetics of anti-tuberculosis drugs (rifampin and levofloxacin pending the participants' drug regimen), to generate ROC at baseline for total area under the concentration curve (AUC). Urine will then be collected via limited sampling strategy at 2 and 6 months after enrollment to determine correlation with the baseline urine sample.
Correlation of serum mass spectrometry to urine colorimetry for peak concentration of anti-tuberculosis drugs | 6 months after enrollment completed
  Urine colorimetry will be compared to conventional serum mass spectrometry for kinetics of anti-tuberculosis drugs (rifampin and levofloxacin pending the participants' drug regimen), to generate ROC at baseline for peak concentration (Cmax). Urine will then be collected via limited sampling strategy at 2 and 6 months after enrollment to determine correlation with the baseline urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Heysell, Principal Investigator — University of Virginia
Locations (1):
- Irkutsk Regional Clinical Tuberculosis Hospital, Irkutsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hodges J, Waldman AL, Koshkina O, Suzdalnitsky A, Schwendinger J, Vitko S, Plenskey A, Plotnikova Y, Moiseeva E, Koshcheyev M, Sebekin S, Zhdanova S, Ogarkov O, Heysell S, Dillingham R. Process evaluation for the adaptation, testing and dissemination of a mobile health platform to support people with HIV and tuberculosis in Irkutsk, Siberia. BMJ Open. 2022 Mar 29;12(3):e054867. doi: 10.1136/bmjopen-2021-054867. PMID 35351714
- [Derived] Hodges J, Zhdanova S, Koshkina O, Suzdalnitsky A, Waldman AL, Schwendinger J, Vitko S, Plenskey A, Plotnikova Y, Moiseeva E, Koshcheyev M, Sebekin S, Ogarkov O, Dillingham R, Heysell S. Implementation of a Mobile Health Strategy to Improve Linkage to and Engagement with HIV Care for People Living with HIV, Tuberculosis, and Substance Use in Irkutsk, Siberia. AIDS Patient Care STDS. 2021 Mar;35(3):84-91. doi: 10.1089/apc.2020.0233. Epub 2021 Feb 3. PMID 33538649